CLINICAL TRIAL: NCT01110993
Title: Prospective, Non-interventional, Multicenter Study to Evaluate QoL and Influence of Cognitive Status on QoL in Patients With RRMS During 2 Years Treatment With RNF
Brief Title: An Observational Study to Evaluate Quality of Life (QoL) and Influence of Cognitive Status on QoL in Patients With Relapsing-Remitting Multiple Sclerosis (RRMS) During 2 Years Treatment With Rebif New Formulation (RNF)
Acronym: MusiClock
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR 701068-516
Record Dates: First submitted 2010-04-06; First posted 2010-04-27 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis, Interferon-beta 1-a
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This is a prospective, non-interventional, multicenter study to evaluate quality of life (QoL) and influence of cognitive status on QoL in subjects with relapsing-remitting multiple sclerosis (RRMS) during two years of treatment with Rebif New Formulation (RNF).

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an acquired demyelinating disease of unclear etiology, occurring mainly in adults. Multiple sclerosis occurs in 30-100 people per 100 000. Usually the disease attacks young adults aged between 20 and 40 years. The peak of this occurrence is in the population of 30-35 year olds.

The main feature of the disease is multifocal (disseminated) injury of the central nervous system. The injury causes various neurological symptoms and signs that go on and off (relapsing-remitting form) or progress steadily, and with time cause irreversible damage of the nervous system and permanent disability. In neuropsychological studies, 40-65% of MS subjects show cognitive impairment with prominent involvement of memory, sustained attention and information processing speed. Multiple sclerosis subjects with different disease courses have different cognitive profiles.

Cognitive dysfunction can have a dramatic impact on a subject's QoL, influencing the fulfillment in work and social life, independently from physical disability. The methodology of cognitive status assessment in MS is based on established sets of tests, which could be conduced by qualified neurophysiologists. There is a need of simple test that could be quickly conducted by every physician, providing information of cognitive status/ or one of its parameters (attention/concentration). That kind of information could be immediately used by the physician during the visit to adjust the way of taking history or giving advices to subjects.

During the last 10 years there's been an enormous progress in the MS treatment. New drugs appeared that proved to diminish clinical activity of the disease and slow its progress. Early treatment with disease modifying therapies may reduce cognitive impairment or slow down the progression of cognitive deficits.

The scope of this study is to evaluate the cognitive status (attention/concentration) and the influence of cognitive impairment on QoL in subjects with RRMS during two years of treatment with RNF.

OBJECTIVES

Primary objective:

* To evaluate the QoL in subjects with RRMS during two years of treatment with RNF

Secondary objectives:

* To evaluate the cognitive status (attention/concentration) and the influence of cognitive impairment on QoL in subjects with RRMS during two years of treatment with RNF Subjects will be treated according to widely-acknowledged standards for MS treatment and the choice of drug will depend solely on medical indications. The potential subjects will have been prescribed Rebif for the first time by their treating physicians and will then be given the option to enter in this observational study. As this is purely an observational study, the subjects will be followed by their treating physicians, according to current medical practice and Rebif SmPC (Summary of Product Characteristics) requirements (i.e monitoring of thyroid and liver enzymes prior to the start of therapy, and hepatic function at months 1, 3, 6 and periodically thereafter, prescription of antipyretics etc.) After each control visit, the treating physician will complete subject's observations chart. The planned schedule of visits will be identical to the routine schedule of control visits dictated by the National Health Found: 1st Visit - 3 months after RNF therapy start, 2nd Visit - after 6 months, 3rd Visit - after 9 months, 4th Visit - after 12 months, 5th Visit - after 18 months, 6th Visit - after 24 months.

"0" visit - doctors will be asked to complete data from subjects history (doctors will be given the proposal of testing (MusiQoL[Multiple Sclerosis International Quality of Life], MMSE [Mini Mental State Examination] and 10-PCT [10-Point Clock Test]) most subjects on the visit when the disease-modifying drugs [DMD] therapy is instituted).

ELIGIBILITY:
There are no specific inclusion/exclusion criteria as the trial is a non-interventional, observational study. The criteria are based on SmPC and criteria of Polish National Found Programme of RRMS Patients Treatment:

Inclusion Criteria:

* Subjects aged above 18 years
* Subjects with clinically diagnosed RRMS which is characterised by two or more acute exacerbations in the previous two years
* Subjects who has never been treated with Rebif (previous treatment with other DMDs will not be regarded as an exclusion criterion)
* Written consent to cooperation made by the environmental nurse who takes care about subject in hospital as well as in his home
* Score of 21 or more points, according to National Heath Found Patient inclusion criteria for the 2 years program of MS treatment with interferon beta

Exclusion Criteria:

Exclusion criteria conform with Rebif's registered contraindications, described in an Sm PC approved by Ministry of Health.

* Interferon beta-1a is contraindicated during pregnancy
* Interferon beta-1a is contraindicated in subjects with confirmed hypersensitivity to natural or recombined interferon beta, or to any of the adjuvant substances
* Interferon beta-1a is contraindicated in subjects with severe depression and/or suicidal thoughts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with Multiple Sclerosis undergoing treatment with Rebif in Poland.
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2010-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Quality of Life | Baseline to 24 months of RNF treatment (At baseline, 12 and 24 months)
  To evaluate the QoL by assessing the changes in MusiQoL Questionaire scores

SECONDARY OUTCOMES:
Assessment of Cognitive Status | Baseline to 24 months of RNF treatment (At baseline, 12 and 24 months)
  To evaluate cognitive status by assessing the changes in MMSE and 10-PCT scores
Influence of cognitive impairment on QoL in subjects with RRMS | Baseline to 24 months of RNF treatment (At baseline, 12 and 24 months)
  To evaluate the influence of cognitive impairment on QoL in subjects with RRMS by assessing the correlation between changes in MusiQoL and those in 10-PCT and MMSE
Assessment of Expanded Disability Status Scale | Baseline to 24 months of RNF treatment (At baseline, 12 and 24 months)
Assessment of number of relapses | Baseline to 24 months of RNF treatment (At baseline, 12 and 24 months)
Assessment of results of Evoked Potentials (visual, auditory, somatosensory/ if they are routinely done) | Baseline to 24 months of RNF treatment (At baseline, 12 and 24 months)
Assessment of Magnetic Resonance Imaging results | Baseline to 24 months of RNF treatment (At baseline, 12 and 24 months)
  MRI results will be assessed to depict new Gd-enhancing lesions, new T2 lesions, enlarging T2 (BOD) lesions, new T1 hypointense lesions, enlarging T1 hypointense lesions, atrophy /if they are routinely done

CONTACTS AND LOCATIONS:
Overall Officials: Zbigniew Stelmasiak, Prof., Principal Investigator — Medical University, Department of Neurology, Lublin, Poland
Locations (1):
- Medical University, Department of Neurology, Lublin, Poland